CLINICAL TRIAL: NCT03958812
Title: The Diagnostic Power of VOCs Compared With CTCs for Cancer
Brief Title: Diagnostic Power Comparison Between VOCs and CTCs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Anhui Medical University (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Principal Investigator, Hu Liu, Associate Professor, Anhui Provincial Hospital
Other Study IDs: DPCVC
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Circulating Tumor Cell; Volatile Organic Chemicals; Breast Cancer; Gastric Cancer; Diagnoses Disease
Keywords: CTCs; VOCs; Breast cancer; Gastric cancer; diagnoses
MeSH Terms: conditions — Neoplastic Cells, Circulating; Breast Neoplasms; Stomach Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Gastric cancer: patients with definitive diagnosis of gastric cancer by pathology
  Interventions: Diagnostic Test: Circulating tumor cells, Volatile organic compounds
- Breast cancer: patients with definitive diagnosis of breast cancer by pathology
  Interventions: Diagnostic Test: Circulating tumor cells, Volatile organic compounds
- Benign gastric diseases: Gastritis or gastric ulcer
  Interventions: Diagnostic Test: Circulating tumor cells, Volatile organic compounds
- Benign breast diseases: Hyperplasia of mammary glands or mastitis
  Interventions: Diagnostic Test: Circulating tumor cells, Volatile organic compounds
- Normal: healthy volunteers
  Interventions: Diagnostic Test: Circulating tumor cells, Volatile organic compounds

INTERVENTIONS:
Diagnostic Test: Circulating tumor cells, Volatile organic compounds — Alveolar exhaled breath samples and peripheral venous blood(10ml) will be collected from each patients

SUMMARY:
Early diagnosis of malignant tumors is pivotal for improving their prognoses. Circulating tumor cells (CTC) in peripheral blood and Volatile organic compounds (VOCs) in exhaled breath are newly developed diagnosis method. Due to the low percentage of CTCs in peripheral blood of cancer patients and the surface structure of lymphocytes (especially megakaryocytes) is often confused with tumor cells, CTC has a high false positive and negative rate. In recent years, the detection of volatile organic compounds (VOCs) in exhaled breath as a simple and noninvasive method has shown broad application prospects in the diagnosis of various diseases. A series of studies of VOCs diagnosing solid tumors the investigators had conducted in the past decade show that VOCs can not only distinguish different types of tumors, but also can make a distinction between different stages. This study was to compare CTC and VOCs with clinical samples. Predictive models will be built employing discriminant factor analysis (DFA) pattern recognition method. Sensitivity and specificity will be determined using leave-one-out cross-validation or an independent blind test set.

DETAILED DESCRIPTION:
200 patients with definitive diagnoses will be enrolled and the alveolar exhaled breath samples and peripheral venous blood will be collected. Two blood samples and two breath samples will be collected from each patient. One blood sample will be send to CTC tests for a blind test and the other will be used for headspace VOCs analyses. One breath sample was used for analysis with the Nano-sensors array, and the other was used for gas chromatography coupled with mass spectrometry (GC-MS) analysis. The VOCs samples were collected using sorbent tubes at a total flow through sorption trap of 200ml/min, then will be send to Israel Institute of Technology for further test.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years
* Definitive diagnosis of gastric cancer, breast cancer,benign breast disease and gastric lesions
* ECOG(Eastern Cooperative Oncology Group) scores ≤ 2

Exclusion Criteria:

* Other palliative chemotherapy and radiotherapy for this cancer
* Other cancer
* Diabetes, Fatty liver
* Autoimmune disease
* Pulmonary ventilation dysfunction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200 patients or volunteers who undergo Gastroscopy or breast surgery in Anhui Provincial cancer hospital, Hefei, China
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-06-15 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Discrimination between Malignant and Benign Gastric/Breast Lesions and normal group with each diagnostic method (Na-nose/GC-MS/CTC) | From June 15,2019 to June 1,2020
  Exhaled breath samples and peripheral venous blood collected will be used to build predictive models employing discriminant factor analysis (DFA) and thereafter examine the sensitivity and specificity of model identification.

SECONDARY OUTCOMES:
Comprehensive diagnostic model of VOCs and CTCs | From June 1,2020 to Dec 31,2020
  Organize predictive models of VOCs/CTCs and establish Comprehensive Diagnostic Model.

CONTACTS AND LOCATIONS:
Overall Officials: Hu Liu, MD, Principal Investigator — Anhui Provincial Cancer Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barash O, Zhang W, Halpern JM, Hua QL, Pan YY, Kayal H, Khoury K, Liu H, Davies MP, Haick H. Differentiation between genetic mutations of breast cancer by breath volatolomics. Oncotarget. 2015 Dec 29;6(42):44864-76. doi: 10.18632/oncotarget.6269. PMID 26540569
- [Background] Amal H, Shi DY, Ionescu R, Zhang W, Hua QL, Pan YY, Tao L, Liu H, Haick H. Assessment of ovarian cancer conditions from exhaled breath. Int J Cancer. 2015 Mar 15;136(6):E614-22. doi: 10.1002/ijc.29166. Epub 2014 Sep 5. PMID 25159530
- [Background] Nakhleh MK, Amal H, Jeries R, Broza YY, Aboud M, Gharra A, Ivgi H, Khatib S, Badarneh S, Har-Shai L, Glass-Marmor L, Lejbkowicz I, Miller A, Badarny S, Winer R, Finberg J, Cohen-Kaminsky S, Perros F, Montani D, Girerd B, Garcia G, Simonneau G, Nakhoul F, Baram S, Salim R, Hakim M, Gruber M, Ronen O, Marshak T, Doweck I, Nativ O, Bahouth Z, Shi DY, Zhang W, Hua QL, Pan YY, Tao L, Liu H, Karban A, Koifman E, Rainis T, Skapars R, Sivins A, Ancans G, Liepniece-Karele I, Kikuste I, Lasina I, Tolmanis I, Johnson D, Millstone SZ, Fulton J, Wells JW, Wilf LH, Humbert M, Leja M, Peled N, Haick H. Diagnosis and Classification of 17 Diseases from 1404 Subjects via Pattern Analysis of Exhaled Molecules. ACS Nano. 2017 Jan 24;11(1):112-125. doi: 10.1021/acsnano.6b04930. Epub 2016 Dec 21. PMID 28000444
- [Background] Leja MA, Liu H, Haick H. Breath testing: the future for digestive cancer detection. Expert Rev Gastroenterol Hepatol. 2013 Jul;7(5):389-91. doi: 10.1586/17474124.2013.811033. No abstract available. PMID 23899275
- [Background] Amal H, Leja M, Broza YY, Tisch U, Funka K, Liepniece-Karele I, Skapars R, Xu ZQ, Liu H, Haick H. Geographical variation in the exhaled volatile organic compounds. J Breath Res. 2013 Dec;7(4):047102. doi: 10.1088/1752-7155/7/4/047102. Epub 2013 Nov 1. PMID 24184568
- [Background] Amal H, Ding L, Liu BB, Tisch U, Xu ZQ, Shi DY, Zhao Y, Chen J, Sun RX, Liu H, Ye SL, Tang ZY, Haick H. The scent fingerprint of hepatocarcinoma: in-vitro metastasis prediction with volatile organic compounds (VOCs). Int J Nanomedicine. 2012;7:4135-46. doi: 10.2147/IJN.S32680. Epub 2012 Jul 30. PMID 22888249